CLINICAL TRIAL: NCT01125163
Title: Randomized Trial Comparing Iron Supplementation Versus Routine Iron Intake in Very Low Birth Weight Infants
Brief Title: Trial Comparing Iron Supplementation Versus Routine Iron Intake in Very Low Birth Weight Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: HSC-MS-10-0031
Record Dates: First submitted 2010-05-13; First posted 2010-05-18 (Estimated); Results first posted 2019-01-04 (Actual); Last update posted 2019-01-04 (Actual); Status verified 2018-07

CONDITIONS: Iron Deficiency Anemia
Keywords: very low birth weight infants; anemia; iron supplementation
MeSH Terms: conditions — Anemia, Iron-Deficiency; Anemia | interventions — Iron-Dextran Complex; Geritol; Iron

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- multivitamin with iron (Active Comparator): daily oral multivitamin providing 2mg/kg of iron
  Interventions: Dietary Supplement: Iron Supplement
- multivitamin without iron (Placebo Comparator): daily oral multivitamin without iron
  Interventions: Dietary Supplement: multivitamin

INTERVENTIONS:
Dietary Supplement: Iron Supplement — multivitamin that provides 2mg/kg/day of iron given orally to infants when they are tolerating 120 ml/dg/day of preterm formula or fortified breast milk until they reach 36 weeks adjusted postmenstrual age.
  Other Names: iron supplementation
  Arms: multivitamin with iron
Dietary Supplement: multivitamin — daily oral multivitamin without iron until 36 weeks adjusted postmenstrual age
  Other Names: Multivitamin without iron
  Arms: multivitamin without iron

SUMMARY:
In preterm infants with birth weights less than 1500 grams, does iron supplementation with 2mg/kg/day in addition to routine feeding with routine iron-fortified milk (formula or fortified mother's milk), as compared to routine iron fortified milk, increase hematocrit at 36 weeks adjusted postmenstrual age (or at discharge if sooner)?

DETAILED DESCRIPTION:
Fortified mother's milk or fortified formula is routine practice in neonatal units and is not an intervention.

ELIGIBILITY:
Inclusion Criteria:

* Birth weight <1500 grams
* Tolerating iron fortified preterm formula or fortified human milk at 120cc/kg/day by 8 weeks of age
* </= 32 weeks adjusted post-menstrual age at the time of enrollment

Exclusion Criteria:

* Cyanotic heart disease
* Bowel resection prior to enrollment

Ages: 24 Weeks to 32 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 150 (Actual)
Dates: Start 2010-05; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tiffany Taylor, M.D., Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- Children's Memorial Hermann Hospital, Texas Medical Center, Houston, Texas, United States

REFERENCES:
- [Derived] Taylor TA, Kennedy KA. Randomized trial of iron supplementation versus routine iron intake in VLBW infants. Pediatrics. 2013 Feb;131(2):e433-8. doi: 10.1542/peds.2012-1822. Epub 2013 Jan 21. PMID 23339225

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Multivitamin With Iron | Multivitamin Without Iron
Started | 76 | 74
Completed | 76 | 74
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Multivitamin With Iron | Multivitamin Without Iron | Total
Number analyzed (Participants) | 76 | 74 | 150
Age, Continuous [Mean (Standard Deviation); unit: gestational age (weeks)] — Infants with birth weight <1500 g who reached 120 ml/kg/day of feedings prior to 32 wks postmenstrual age were eligible.
  gestational age (weeks) | 27.3 (2.0) | 27.3 (2.1) | 27.3 (2)
Sex: Female, Male [Count of Participants; unit: Participants] — number of females and males per group (intervention and control)
  Participants
    Female | 38 | 35 | 73
    Male | 38 | 39 | 77
Region of Enrollment [Number; unit: participants]
  United States | 76 | 74 | 150

OUTCOME MEASURES:

1. Primary Outcome: Hematocrit (Hct) at 36 Wks Post Menstrual Age (PMA)
Description: For infants discharged home prior to 36 wks PMA, the last Hct was used.For infants transferred prior to 36 wks PMA, the Hct at receiving hospital was used if available. A non-parametric rank sum analysis was performed as follows so that infants who died before 36 wks and those transfused could be included in an intention-to-treat analysis.Infants were ranked by death (lowest rank) then by number of transfusions (next lowest ranks). For infants who survived and were not transfused, the 36 wk PMA Hct was used as the primary outcome.
Time Frame: at 36 weeks adjusted postmenstrual age
Population: Sample size was based on a retrospective observational pilot study from the 2008 calendar year. A sample size of 75 per group was chosen to achieve 80% power to detect a difference in Hct of 2 % between groups, assuming a mean Hct of 25.6% in the control group, a standard deviation 4.4%, with alpha level (0.05) using a two-sided two-sample t-test.
Measure: Mean (Standard Deviation); unit: % Hematocrit
Groups:
- Multivitamin With Iron: daily oral multivitamin providing 2mg/kg/day of iron
Arm/Group | Multivitamin With Iron | Multivitamin Without Iron
Number analyzed (Participants) | 76 | 74
% Hematocrit | 29.2 (4.0) | 28.2 (4.5)
Statistical Analysis 1: Comparison: Multivitamin With Iron vs Multivitamin Without Iron; A non-parametric rank sum analysis was performed as follows so that infants who died before 36 wks and infants who were transfused could be included in an intention-to-treat analysis. Infants were ranked by death (lowest rank) then by number of transfusions (next lowest ranks). For infants who survived and were not transfused, the 36 wks PMA Hct was used as the primary outcome; Test type: Superiority or Other; p = 0.59, Wilcoxon (Mann-Whitney) — All infants were analyzed according to their assigned groups

2. Secondary Outcome: Number of Participants Who Received Red Cell Transfusions During Intervention Period
Description: The numbers below represent the number of participants in each arm that received a transfusion during intervention period.
Time Frame: from study day 1 to 36 week adjusted postmenstrual age or discharge if the infant is discharged sooner
Measure: Number; unit: participants
Arm/Group | Multivitamin With Iron | Multivitamin Without Iron
Number analyzed (Participants) | 76 | 74
participants | 48 | 54
Statistical Analysis 1: Comparison: Multivitamin With Iron vs Multivitamin Without Iron; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.64, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Arm/Group | Multivitamin With Iron | Multivitamin Without Iron
Serious Adverse Events (participants affected / at risk) | 1/76 | 1/74
Other Adverse Events (participants affected / at risk) | 0/76 | 0/74
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Multivitamin With Iron (N=76) | Multivitamin Without Iron (N=74)
Death (Gastrointestinal disorders) | 1/13 (1) | 1/9 (1) — The two infants (one in each group) died of Necrotizing Entercolitis which is an illness that occurs in extremely premature infants.

LIMITATIONS AND CAVEATS:
This trial was done in a setting where relatively liberal transfusion guidelines (based on PINT study) are used so difficult to generalize to settings where restrictive transfusion guidelines are used.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No